CLINICAL TRIAL: NCT00771381
Title: A Phase II Pre-Treatment Hypoxia PET Imaging Study Using 18F-FAZA in Patients With Invasive Duct Carcinoma of the Breast
Brief Title: A Study to Determine the Value of 18F-FAZA PET Imaging in Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Retirement of former Qualified Investigator and lack of resources to complete study
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KT-FAZ-004
Record Dates: First submitted 2008-09-19; First posted 2008-10-13 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-02

CONDITIONS: Breast Neoplasm
Keywords: 18F-FAZA; 18F-FDG; Positron Emission Tomography; Cell Hypoxia
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 18F-FAZA + FluGlucoScan Injection
  Interventions: Drug: 18F-FAZA PET scan; Drug: FluGlucoScan Injection (18F-FDB) PET scan

INTERVENTIONS:
Drug: 18F-FAZA PET scan — Radioactive dose of 18F-FAZA: 110-600 MBq per injection. One pre-treatment injection of 18F-FAZA and PET scan will be permitted per patient.
Drug: FluGlucoScan Injection (18F-FDB) PET scan — Radioactive dose of 100-700 MBq per injection. A single pre-treatment injection of FluGlucoScan Injection and PET scan will be permitted per patient.

SUMMARY:
In about half the cases of breast cancer, there is hypoxic (no, or little oxygen) tissue present. Hypoxic cells can be resistant to treatment and may cause increased tumour growth. This study will use 18F-FAZA PET scans before surgery or treatment to assess whether patients have hypoxic tumours. The results will be compared to tissue samples removed during surgery and to the distribution of 18F-FDG.

DETAILED DESCRIPTION:
Hypoxia or anoxia can be found in 50% of locally advanced breast carcinomas. Assessment of pre-treatment in viva and in vitro hypoxia could allow patient selection for more aggressive therapy or clinical trails focused on targeting hypoxia. We will use the PET radiotracer 18F-FAZA to monitor hypoxia in the protocol. We will study pathological characteristics on the final tumour restriction specimen and correlate prognostic and predictive factors with PET scan data. Tumour banking is optional.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 years of age. If female of child bearing potential and if outside of the window of 10 days since the first day of the 0last menstrual period, patient will be required to have a negative pregnancy test.
2. Pathologically proven invasive duct carcinoma of the breast (FNA or core biopsy), T1-T4(T ≥ 1.5 cm)
3. FluGlucoScan Injection and 18F-FAZA PET scans performed prior to treatment.
4. FluGlucoScan Injection and 18F-FAZA PET scans performed within 4 weeks prior to their definitive surgery if subject does not have neoadjuvant therapy.
5. Able and willing to follow instructions and comply with the protocol
6. Provide written informed consent prior to participation in the study.
7. ECOG performance score ≤ 2

Exclusion Criteria:

1. Previous malignancy or diagnosis less than ten (10) years ago. Skin Cancers (excluding malignant melanoma) and carcinoma in situ of the cervix are exceptions.
2. Excisional biopsy of the primary breast tumour has been performed
3. Women with an invasive carcinoma of the breast that is not predominantly of the invasive duct subtype
4. Primary breast carcinoma previously treated.
5. Women who are nursing or pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-11-28 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Uptake of 18F-FAZA (RUS and T/B) and its correlation to tumour size, auxiliary nodal status, tumour grade, EP/PR, and HER-2 status, Ki-67, Androgen receptor status (AR), vimentin and basal keratins, HIF-1 a and glomeruloid microvascular proliferation. | 5 years

SECONDARY OUTCOMES:
General biodistribution of 18F-FAZA and FluGlucoScan Injection | 5 years
Comparison of pre-operative 18F-FAZA and FluGlucoScan Injection PET images | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel W Hudson, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada